CLINICAL TRIAL: NCT02379897
Title: Diet, Obesity and Cardiovascular Risk Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Susan Roberts, Senior Scientist, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: R01HL 57981
Record Dates: First submitted 2015-02-14; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Cardiovascular Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Obesity | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- LowGI+ModCarb (Experimental): Low glycemic index + moderate carbohydrate/moderate fat diet
  Interventions: Other: Diet
- LowGI+HighCarb (Experimental): Low glycemic index + high carbohydrate/low fat diet
  Interventions: Other: Diet
- HighGI+ModCarb (Experimental): High glycemic index + moderate carbohydrate/moderate fat diet
  Interventions: Other: Diet
- HighGI+HighCarb (Experimental): High glycemic index + high carbohydrate/low fat diet
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet

SUMMARY:
Controversy exists about the role of dietary glycemic index (GI) and fat content and cardiovascular risk. Our aim was to assess the long term effects of altering dietary GI, carbohydrate, and fat on body weight, lipids, glucose homeostasis, and C reactive protein (CRP) in overweight and obese subjects. Men and post-menopausal women with body mass index values between 28-38 kg/m2 were placed on an isoweight average American diet for 5 weeks, then randomized to one of 4 diets which differed in GI, carbohydrate and fat content with calorie restriction for 12 weeks. The same diets were continued for 5 weeks under isoweight conditions, and in the free-living state for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI 28-28 kg/m2
* Male or postmenopausal female 45-65 yr

Exclusion Criteria:

* Abnormal thyroid, liver, kidney function
* Abnormal hemoglobin
* LDL-cholesterol ≤ 100 mg/dL
* Fasting triglycerides ≥ 400 mg/dL
* Diabetes or on medication for diabetes
* Chronic illness
* Elevated blood lipids

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2000-09; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline to 12 weeks

SECONDARY OUTCOMES:
Change in fasting plasma high density lipoprotein cholesterol | Baseline to 12 weeks, 17 weeks, and 16 months
Change in fasting plasma low density lipoprotein cholesterol-cholesterol | Baseline to 12 weeks, 17 weeks, and 16 months
Change in fasting plasma very low density lipoprotein cholesterol-cholesterol | Baseline to 12 weeks, 17 weeks, and 16 months
Change in fasting plasma triglycerides | Baseline to 12 weeks, 17 weeks, and 16 months
Change in fasting plasma insulin | Baseline to 12 weeks, 17 weeks, and 16 months
Change in fasting blood glucose | Baseline to 12 weeks, 17 weeks, and 16 months
Change in glycated hemoglobin | Baseline to 12 weeks, 17 weeks, and 16 months
Change in plasma C-reactive protein | Baseline to 12 weeks, 17 weeks, and 16 months
Change in body fat | Baseline to 12 weeks and 17 weeks
Change in resting metabolic rate | Baseline to 12 weeks and 17 weeks
Change in blood pressure | Baseline to 12weeks, 17weeks and 16months
Change in body weight | Baseline to 17weeks and 16months
Change in postprandial blood glucose | Baseline to 12weeks and 17weeks
  Oral glucose tolerance test